CLINICAL TRIAL: NCT06582186
Title: Individualization of First Maintenance Doses of Voriconazole Using a Multiparametric Algorithm in Hematology Patients: a Prospective Single-arm Interventional Study
Brief Title: Individualized First Maintenance Doses of Voriconazole Through a Multiparametric Algorithm
Acronym: VORIPRECI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC23.0230; 2024-A01425-42 (Other: ID RCB)
Record Dates: First submitted 2024-08-22; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Aspergillosis Invasive; Fungal Infection; Hematologic Malignancy
Keywords: model-informed precision dosing; single-arm prospective interventional study; Simon design
MeSH Terms: conditions — Mycoses; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- individualized maintenance doses (Experimental): Individualization of first maintenance doses through a multiparametric algorithm integrating CYP2C19 genotype, C reactive protein level and age
  Interventions: Drug: Individualization of first voriconazole maintenance doses

INTERVENTIONS:
Drug: Individualization of first voriconazole maintenance doses — Individualization of first voriconazole maintenance doses

SUMMARY:
The goal of this interventional single-arm study is to evaluate the interest of a multiparametric algorithm for individualization of first voriconazole maintenance doses for improvement of initial voriconazole exposure in adult patients with haematological malignancies. The main objective it aims is to determine the percentage of patients with initial voriconazole trough concentrations in the therapeutic range after individualization of first maintenance doses.

Participants will benefited from individualization of first voriconazole maintenance doses through a previously developed and validated multiparametric algorithm (publication in progress) taking into account CYP2C19 genotype, C reactive protein level and age.

DETAILED DESCRIPTION:
The currently recommended therapeutic drug monitoring of voriconazole has improved the efficacy of this treatment and reduced its adverse effects, especially for treatment and prophylaxis of invasive aspergillosis. However, dose adjustments made as part of this therapeutic drug monitoring only occur at the earliest 3 to 5 days after the initiation of treatment, whereas it is essential to achieve effective concentrations from the start of treatment. Simple a priori dose adjustment approaches based on CYP2C19 genotype have been shown to improve voriconazole exposure and treatment response. However other factors such as the patient's inflammatory status or age also influence voriconazole exposure, suggesting that strategies for individualizing initial voriconazole doses could be improved by integrating all covariates influencing voriconazole pharmacokinetics. In this line, a previous multicenter and international study has developped and validated an algorithm for calculating the first maintenance doses integrating not only the CYP2C19 genotype, but also the inflammatory status, the patient's age, and the presence (or not) of hematological malignancy. Here, the investigators propose to evaluate the interest of this multiparametric algorithm for improving initial exposure (within the first 4 days) to voriconazole in patients suffering from haematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* adult patient suffering from haematological malignancy
* followed in the clinical hematology department or in the hematology day hospital of the Grenoble Alps University Hospital
* consenting to carrying out CYP2C19 genotyping
* likely to start treatment with voriconazole (for curative or prophylactic purposes as part of care)
* having signed a written consent to participate
* affiliated to a social security system

Exclusion Criteria:

* comedication with strong inhibitors/inducers (valproic acid, phenytoin, carbamazepine, rifampicin)
* Subject during exclusion period from another study,
* Persons referred to in articles L1121-5 to L1121-8 of the CSP (corresponds to all protected persons: pregnant woman, parturient woman, breastfeeding mother, person deprived of liberty by judicial or administrative decision, persons subject to care psychiatric pursuant to articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of article L. 1121-8, persons admitted to a health or social establishment for purposes other than research , minors, person subject to a legal protection measure or unable to express their consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with initial plasma voriconazole trough concentration in the therapeutic range | Day 5 +/-2

SECONDARY OUTCOMES:
Frequency of initial plasma voriconazole trough concentrations above the therapeutic range | Day 5 +/-2
Frequency of initial plasma voriconazole trough concentrations below the therapeutic range | Day 5 +/-2
Voriconazole area under the curve (AUC0-12h) after the first maintenance dose individualized | Day 2
Time to get the therapeutic range | through study completion, an average of 3 months
Treatment outcome in patients curatively treated | At month 3 +/- 15 days
Frequency of side effects | through study completion, an average of 3 months
Percentage of patients with initial plasma voriconazole trough concentration in the therapeutic range | Day 5 +/-2
  comparison with an historic cohort

CONTACTS AND LOCATIONS:
Overall Officials: Gautier-Veyret Elodie, Principal Investigator — Grenoble Alps University Hospital
Locations (1):
- Gautier-Veyret, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gautier-Veyret E, Thiebaut-Bertrand A, Roustit M, Bolcato L, Depeisses J, Schacherer M, Schummer G, Fonrose X, Stanke-Labesque F. Optimization of voriconazole therapy for treatment of invasive aspergillosis: Pharmacogenomics and inflammatory status need to be evaluated. Br J Clin Pharmacol. 2021 Jun;87(6):2534-2541. doi: 10.1111/bcp.14661. Epub 2020 Dec 13. PMID 33217017
- [Background] Bolcato L, Khouri C, Veringa A, Alffenaar JWC, Yamada T, Naito T, Lamoureux F, Fonrose X, Stanke-Labesque F, Gautier-Veyret E. Combined Impact of Inflammation and Pharmacogenomic Variants on Voriconazole Trough Concentrations: A Meta-Analysis of Individual Data. J Clin Med. 2021 May 13;10(10):2089. doi: 10.3390/jcm10102089. PMID 34068031